CLINICAL TRIAL: NCT01539993
Title: Prospective Analysis of Liver Cancer Treatment and Interventions
Brief Title: Prospective Liver Study
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Hyun Kevin Kim, MD FSIR, Director of Interventional Radiology and Image-Guided Medicine., Emory University
Other Study IDs: IRB00014768
Record Dates: First submitted 2012-02-15; First posted 2012-02-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Liver Cancer
Keywords: Hepatocellular carcinoma; Liver metastases; Cholangiocarcinoma; Percutaneous treatments; RFA; TACE; DEB
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This study is designed for patients diagnosed with Liver cancer to collect information about the relationship between types of liver cancer, methods of treatment and outcomes over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Hepatocellular carcinoma and referred for percutaneous liver treatment.

Exclusion Criteria:

* Severe liver disfunction
* Active uncontrolled infection
* Significant underlying medical of physical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 yrs and older with a diagnosis of Hepatocellular carcinoma and elegible for percutaneous liver treatments
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2008-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Assess efficacy of percutaneous and transarterial treatments for liver cancer. | 1 month
  QOL questionnaire will be collected during follow up visit.

SECONDARY OUTCOMES:
long term follow up | 3 months, 6 months 1year
  Patients will be administered QOL during 3 months, 6 months and 1 year follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin S Kim, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States